CLINICAL TRIAL: NCT06902363
Title: Sweat Testing in Infants: a Comparative Study Investigating the Collection of Sweat on the Upper Limbs Compared to the Lower Limbs
Brief Title: Sweat Testing in Infants: Comparing Sweat Collection on Upper Vs Lower Limbs
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: EliTechGroup (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 24147_Zweetteststudi
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Cystic Fibrosis (CF)
Keywords: Cystic fibrosis; Sweat testing; Sweat test; Infants; Quantity non sufficient
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Comparison of Sweat Collection Sites: Forearm vs. Thigh (Experimental): All enrolled infants undergo sweat testing using the Macroduct Advanced device, with simultaneous collection on the forearm (standard site) and thigh (alternative site). The goal is to compare sweat volume and chloride concentration between both anatomical sites, focusing on the rate of quantity not sufficient (QNS) outcomes.
  Interventions: Device: Macroduct Advanced

INTERVENTIONS:
Device: Macroduct Advanced — Sweat stimulation and collection using the Macroduct Advanced system on two anatomical sites (forearm and thigh) in infants under 6 months of age.

SUMMARY:
The goal of this study is to compare the rate of Quantity Not Sufficient (QNS) during sweat collection in infants under 6 months of age, using the Macroduct Advanced device for sweat testing. The main question it aims to answer is:

Does sweat collection from the thigh (lower limb) reduce the QNS rate compared to the forearm (upper limb) in infants? Do chloride concentration levels differ between sweat collected from the forearm and thigh in the same infants?

DETAILED DESCRIPTION:
This is a prospective, observational study aimed at evaluating the effectiveness of the Macroduct Advanced device for sweat testing in infants under 6 months of age. The primary goal is to compare the rate of Quantity Not Sufficient (QNS) between two sweat collection sites: the forearm (upper limb) and the thigh (lower limb). The study seeks to determine whether using the thigh as an alternative collection site can reduce the incidence of QNS, a common challenge in sweat testing in infants, where at least 15 microliters of sweat are required for an accurate result.

Study Objectives:

To assess if sweat collection from the thigh results in a lower QNS rate compared to the forearm in infants.

To compare the chloride concentration levels of sweat collected from both the forearm and thigh, in order to evaluate if the collection site affects the chloride measurements.

Study Design:

Participants will undergo sweat collection from both the forearm and thigh, within the same study session, using the Macroduct Advanced device.

The QNS rate will be recorded for each collection site. Chloride levels from the sweat samples will be measured for comparison between the two sites.

The study will involve healthy infants under 6 months of age, and data will be collected to evaluate the feasibility and effectiveness of using the thigh as a collection site for sweat testing.

Primary and Secondary Outcomes:

Primary Outcome: Reduction in the QNS rate when sweat is collected from the thigh compared to the forearm.

Secondary Outcome: Comparison of chloride concentration levels from the forearm and thigh to determine if there is a significant difference in chloride levels depending on the collection site.

This study will provide valuable insights into improving the accuracy and feasibility of sweat testing in infants, especially in cases where QNS is common and may require repeated tests. If successful, using the thigh as a collection site could enhance the overall success rate of sweat tests and reduce the need for retesting, improving clinical care for infants with conditions such as cystic fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* minimal 3,000 kg
* after a positive newborn screening (NBS) test. During this test, newborns are screened for rare diseases including CF. In case of a positive NBS test for CF, a sweat test is routinely performed to confirm or withdraw the diagnosis.
* after clinical assessment for CF, with ST as diagnostic step
* siblings of patients with CF in order to exclude CF
* CF patients who are willing to participate
* Healthy infants, born at the maternity unit of UZ Brussel, of which parents are willing to participate

Exclusion Criteria:

* chromosome abnormalities
* metabolic abnormalities
* cardiopathies
* eczema
* important skin lesions on the limbs
* use of systemic corticosteroids
* critically ill patients (for example hemodynamically unstable)

Ages: 10 Days to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-03-30 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of Sweat Collection Sites: Forearm vs. Thigh in Infants (Primary Outcome: QNS Rate) | Measurement of QNS rate will be taken at the time of sweat collection from both forearm and thigh, during each testing session. Data will be recorded in real-time, and analysis will occur immediately following the collection.
  The primary objective of this study is to compare the rate of Quantity Not Sufficient (QNS) between sweat collected from the forearm (upper limb) and the thigh (lower limb) in infants under 6 months of age. Both sites will be tested on the same infant at the same time using the Macroduct Advanced device. The goal is to determine whether sweat collection from the thigh reduces the incidence of QNS compared to the forearm, which is the traditional site for sweat testing in infants. Additionally, the study aims to assess if the circumferential size of the upper and lower limbs influences the rate of QNS.

SECONDARY OUTCOMES:
Comparison of Chloride Concentration between Forearm and Thigh Sweat Collection in Infants | Chloride concentration will be measured immediately after sweat collection from both forearm and thigh during each session, with results recorded and analyzed following each collection.
  The secondary objective of this study is to compare chloride concentration values between sweat collected from the forearm (upper limb) and the thigh (lower limb) in the same infant under 6 months of age. Sweat will be collected simultaneously from both sites using the Macroduct Advanced device. This comparison aims to determine if there is a significant difference in chloride levels between the two sites, and whether the anatomical site of sweat collection impacts the chloride concentration in the samples.

CONTACTS AND LOCATIONS:
Overall Officials: Elke De Wachter, Prof. Dr., Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- UZ Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McColley SA, Elbert A, Wu R, Ren CL, Sontag MK, LeGrys VA. Quantity not sufficient rates and delays in sweat testing in US infants with cystic fibrosis. Pediatr Pulmonol. 2020 Nov;55(11):3053-3056. doi: 10.1002/ppul.25027. Epub 2020 Aug 25. PMID 32797669
- [Background] Taylor NA, Machado-Moreira CA. Regional variations in transepidermal water loss, eccrine sweat gland density, sweat secretion rates and electrolyte composition in resting and exercising humans. Extrem Physiol Med. 2013 Feb 1;2(1):4. doi: 10.1186/2046-7648-2-4. PMID 23849497
- [Background] Vermeulen F, Lebecque P, De Boeck K, Leal T. Biological variability of the sweat chloride in diagnostic sweat tests: A retrospective analysis. J Cyst Fibros. 2017 Jan;16(1):30-35. doi: 10.1016/j.jcf.2016.11.008. Epub 2016 Dec 22. PMID 28017620
- [Background] Massie J, Greaves R, Metz M, Wiley V, Graham P, Shepherd S, Mackay R. Australasian Guideline (2nd Edition): an Annex to the CLSI and UK Guidelines for the Performance of the Sweat Test for the Diagnosis of Cystic Fibrosis. Clin Biochem Rev. 2017 Nov;38(3):115-130. No abstract available. PMID 29332976
- [Background] LeGrys VA, Briscoe D, McColley SA. Sweat testing: specimen collection and quantitative chloride analysis. CLSI Guideline 2019;C34
- [Background] Cirilli N, Southern KW, Barben J, Vermeulen F, Munck A, Wilschanski M, Nguyen-Khoa T, Aralica M, Simmonds NJ, De Wachter E; ECFS Diagnostic Network Working Group. Standards of care guidance for sweat testing; phase two of the ECFS quality improvement programme. J Cyst Fibros. 2022 May;21(3):434-441. doi: 10.1016/j.jcf.2022.01.004. Epub 2022 Jan 19. PMID 35063396
- See also: Classification of people based on ethnicity — https://grants.nih.gov/grants/guide/notice-files/NOT-OD-15-089.html